CLINICAL TRIAL: NCT02197702
Title: Vitamin D In the Prevention of Viral-induced Asthma of Preschoolers: a Randomised Controlled Trial (RCT)- (DIVA)
Brief Title: Vitamin D in Preschoolers With Viral-induced Asthma
Acronym: DIVA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Montreal Children's Hospital of the MUHC (Other); British Columbia Children's Hospital (Other); London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Professor Francine Ducharme, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DIVA
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: RCT; asthma; pediatric; virus; corticosteroid
MeSH Terms: conditions — Asthma; Virus Diseases | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: identical placebo
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 ml identical placebo taken by mouth at baseline and 3.5 months.
  Interventions: Dietary Supplement: placebo
- Vitamin D (Experimental): Vitamin D (100,000IU) given in a 2 ml oral dose at baseline and 3.5months.
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — Two doses of cholecalciferol 100,000 unit (2 mL) given 3.5 months apart, once in the fall, once in the winter
  Other Names: cholecalciferol
  Arms: Vitamin D
Dietary Supplement: placebo — Two doses of identical placebo (2 mL) given 3.5 months part, once in the fall, once in the winter
  Arms: Placebo

SUMMARY:
In this 7-month randomized controlled trial, children aged 1-6 years with asthma attacks triggered mostly by colds, will receive a high dose of vitamin D or a placebo every 3.5 months during their usual clinic visit. This study will test whether children receiving a high dose of vitamin D have less frequent and less severe asthma exacerbations compared with those receiving placebo.The study will also document the safety profile of this strategy.

DETAILED DESCRIPTION:
IMPORTANT NOTE: Due to receiving a 2-year partial funding enabling only a single-centre pilot trial, rather than an adequately-powered multicentre study, the primary outcome was modified post hoc for the overall change from baseline in total serum 25OHD during the study as well as at 3.5 and 7 months, similar to our previous pilot study.(NCT01999907) Post hoc secondary outcomes included the group difference in the proportion of children with total 25OHD ≥75 nmol/L at 3.5 and 7 months and in the rate of oral corticosteroid courses per child. Other a priory specified outcomes included the proportion of children with hypercalciuria (Ca:Cr) >1.25 (1-2 years), >1 (2-5 years) nmol/nmol at any point in time; proportion of children with ≥1 exacerbation requiring rescue oral steroids (former primary outcome); number of emergency department (ED) visits; intensity and duration of asthma symptoms and cumulative use of rescue ß2-agonist use, documented on Asthma Flare-up Diary for Young Children (ADYC); the impact of parents' functional status during exacerbations ascertained on the Effect of a child's asthma flare-up on parents; and duration of URTI.

Based on this analysis of this new post-hoc primary outcome, we have changed the intervention and the primary outcome and obtained funding for a new large multicentre study NCT03365687. it is thus important to share the results of this current trial with other investigators

PRIOR REPORTED DESCRIPTION Design: A multicenter triple-blind randomized parallel-group, placebo-controlled trial of vitamin D3 supplementation. Children aged 1-5 years with (i) physician-diagnosed asthma, predominantly triggered by upper respiratory tract infections (URTIs), (ii) ≥4 reported URTIs in the past year, and (iii) ≥1 exacerbation requiring OCS (a recognised marker of moderate and severe exacerbations) in the past 6 months or ≥2 in the past 12 months, will be randomly allocated to one of two treatments in blocks of 4-6, stratified on recruitment site: Intervention group (n=432)-100,000 IU oral vitamin D3; control group (n=432)-identical placebo, for 2 oral doses, 3.5 months apart. Co-intervention with asthma therapy (preventive or pre-emptive ICS) will be left to the discretion of the physician and documented. Children will be followed every 3.5 months as per usual practice, with a home visit 10 days after each bolus, during which urine and blood will be sampled for urinary calcium:creatinine ratio, serum vitamin D, markers of calcium metabolism, and mechanistic exploration. A validated diary will serve to document the intensity and severity of exacerbations. In two sites, preschool lung function will be documented (if ≥ 3yrs). Outcomes: Primary endpoint-number of exacerbations requiring rescue oral corticosteroids (OCS) per child, documented by medical and pharmacy records. Secondary outcomes: duration and severity of exacerbations (symptoms & β2-agonist use, by diary; emergency visits, by medical records), parental functional status (by validated instrument), asthma therapy intensification and health care and direct costs (by health records & parent reports). Safety, mechanistic, exploratory outcomes: hypercalciuria, calcium metabolism, excess vitamin D, change in serum gene expression at 10 days (first 25 patients); and change from baseline at 7 months in preschool lung function (2 sites). Based on 3 published RCTs, a sample of 432 per arm (400+7.5% attrition) will provide 80% power (2-tailed alpha of 5%) to detect a 25% reduction in number of exacerbations requiring OCS/child (0.55 vs. 0.4125).

ELIGIBILITY:
Inclusion Criteria:

* age 1-5 years
* physician-diagnosed asthma as per the Global Initiative for Asthma (GINA) guidelines
* URTIs as the main asthma trigger (parental report)
* ≥4 URTIs in the past 12 months (parental report)
* ≥1 asthma exacerbation requiring rescue oral corticosteroids (OCS) in the past 6 months or ≥2 in the past 12 months

Exclusion Criteria:

* intake or intention to use more than 400 IU/day of vitamin D supplement
* extreme prematurity (<28 weeks gestation)
* infants <12 months of age
* no vitamin D supplementation when breast-fed
* recent (<1 year) immigrants from a region at high risk of rickets
* children with vitamin D restrictive diets e.g. vegans
* other chronic respiratory disease (broncho-pulmonary dysplasia; cystic fibrosis)
* condition(s) that alter calcium or vitamin D metabolism/absorption (hypo/hyperparathyroidism, kidney/liver disease, inflammatory bowel disease)
* medications that interfere with vitamin D metabolism (anti-epileptics, diuretics, antacids, anti-fungal drug)
* vitamin D supplementation >1000 IU/ day in last 3 months
* anticipated difficult follow-up (unable to attend clinic visits; plan to leave the province).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ducharme FM, Jensen M, Mailhot G, Alos N, White J, Rousseau E, Tse SM, Khamessan A, Vinet B. Impact of two oral doses of 100,000 IU of vitamin D3 in preschoolers with viral-induced asthma: a pilot randomised controlled trial. Trials. 2019 Feb 18;20(1):138. doi: 10.1186/s13063-019-3184-z. PMID 30777118
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- See also: article — http://pubmed.ncbi.nlm.nih.gov/30777118/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 24 | 23
Withdrew at Visit 1 | 0 | 1
Withdrew at Visit 2 | 1 | 1
Withdrew at Visit 3 | 0 | 2
Analysed for Main Outcome | 23 | 22
Completed | 23 | 19
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.9 (1.2) | 2.9 (0.9) | 2.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 14 | 16 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 16 | 12 | 28
  Ethnicity: Other | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 23 | 47
Vitamin D intake IU/day -Median (25%, 75%) [Median (Inter-Quartile Range); unit: IU/day] | 238 [162 to 270] | 182 [125 to 425] | 215 [165 to 356]
Serum vitamin D <75 nmol/L - n (%) [Count of Participants; unit: Participants] | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum 25OHD
Description: Group difference in the adjusted change from baseline 25OHD over 7 months
Time Frame: During the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 23 | 22
nmol/L | 4.3 [-6.6 to 15.1] | 9.6 [-6.6 to 19.6]

2. Secondary Outcome: Number of Participants With Total 25OHD ≥75 Nmol/L
Description: Group difference in the number of participants with total 25OHD ≥75 nmol/L
Time Frame: at 3.5 and 7 months
Population: The numbers of participants analyzed in Placebo and Vitamin D groups were 23 and 19 at 3.5 months time point, and 22 and 18 at 7 months time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 23 | 19
Participants
  at 3.5 months | 9 | 12
  at 7 months: number analyzed (Participants) | 22 | 18
  at 7 months | 8 | 10

3. Secondary Outcome: Emergency Department Visit for an Asthma Flare-up
Description: Group difference in the number of emergency department visits for asthma per child
Time Frame: During the 7-month follow-up period
Population: The numbers of participants analyzed were 24 in Placebo and 23 in Vitamine D groups.
Measure: Mean (95% Confidence Interval); unit: visits/child
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
visits/child | 1.00 [0.67 to 1.49] | 1.04 [0.70 to 1.56]

4. Other Pre Specified Outcome: Hypercalciuria
Description: Group difference in the number of participants with ≥1 occurrence of hypercalciuria (urinary calcium: creatinine greater than 1.25mmol/mmol for children aged 1-2yrs or greater than 1mmol/mmol for those aged 2-5yrs)
Time Frame: At any point during the 7-month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Participants | 8 | 4

5. Other Pre Specified Outcome: Elevated Serum 25-hydroxyvitamin D (25OHD)
Description: Number of Participants with ≥1 occurrence of elevated serum 25OHD (greater than 225 nmol/L)
Time Frame: At any point during the 7-month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Participants | 0 | 6

6. Other Pre Specified Outcome: Perturbation of the Calcium Homeostasis
Description: Number of participants with ≥1 occurrence of a clinically significant perturbation of the calcium homeostasis (serum Ca, Ph, Alkaline phosphatase), defined as outside normal laboratory values
Time Frame: At any point during the 7-month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of URTIs (Verbal Report)
Description: Adjusted Incidence proportion of URTIs (the event rate per child occurring during the 7-month follow up period)
Time Frame: During the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: number of URTI/child
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 22 | 22
number of URTI/child | 4.12 [3.37 to 5.03] | 4.48 [3.66 to 5.49]

8. Other Pre Specified Outcome: Viral Upper Respiratory Tract Infections (URTI)
Description: Group difference in the number of reported viral upper respiratory tract infections reported in the ADYC diary.
Time Frame: During the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: Viral URTI/child
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Viral URTI/child | 4.24 [3.32 to 5.42] | 3.63 [2.7 to 4.87]

9. Other Pre Specified Outcome: Rescue β2-agonist Use During an Asthma Flare-up (Standardized Over 7 Days)
Description: Group difference in the cumulative daily use of rescue β2-agonist use, standardized over 1 week, as documented by parents on the 'Asthma Flare-up Diary for Young CHildren' (ADYCs) during a URTI or an asthma exacerbation. A cumulative number of inhalations documented in ADYC were divided by the number of days of asthma exacerbation and multiplied by 7 days. Albuterol doses received during acute care visits and hospital admissions were not considered.
Time Frame: During the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: cumulative number of puffs standardized
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
cumulative number of puffs standardized | 41.2 [32.1 to 50.2] | 40.1 [30.4 to 49.8]

10. Other Pre Specified Outcome: Severity of Asthma Symptoms During an Asthma Flare-up (Cumulative Daily Score Standardized Over 7 Days)
Description: Group difference in the severity on the asthma symptoms documented as the sum of daily score on the 'Asthma FLare-up DIary for Young Children' questionnaire where best =1, worst = 7 on each day during asthma flare-up. Since the flare-up typically lasts several days, the cumulative daily score, standarized over 7 days (total possible scale range: 7-49), may increase due to severity or due to the duration of the event. Lower scores indicate lowest severity, higher score indicate longer or higher severity of symptoms.
Time Frame: During an URTI or flare-up during the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: score on a ADYC scale
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
score on a ADYC scale | 12.5 [9.8 to 15.1] | 11.0 [8.9 to 13.2]

11. Other Pre Specified Outcome: Duration of Asthma Symptoms During a Flare-up (by Diary)
Description: Group difference in the duration of asthma symptoms documented on the 'Asthma FLare-up DIary for Young Children' questionnaire
Time Frame: During an URTI or flare-up during the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: days/exacerbation
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
days/exacerbation | 5.2 [4.2 to 6.2] | 5.1 [3.1 to 7.0]

12. Other Pre Specified Outcome: Number of Asthma Exacerbations/Child
Description: The number of asthma exacerbations requiring rescue oral corticosteroids per child
Time Frame: During the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: Courses of oral steroids/child
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Courses of oral steroids/child | 0.79 [0.51 to 1.24] | 0.96 [0.63 to 1.45]

13. Other Pre Specified Outcome: Impact of Exacerbations on Caregivers' Functional Status
Description: Group difference in the caregivers' functional status measured on the 'Effect of a child's asthma flare-up on parents' (ECAP) questionnaire (best =7, worst = 1)
Time Frame: During an URTI or flare-up during the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: Score of a scale
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
Score of a scale | 3.2 [2.6 to 3.8] | 3.3 [2.8 to 3.9]

14. Other Pre Specified Outcome: Caregivers' Workday Lost (in Days Per Flare-up)
Description: Mean group difference in the caregivers' number of workdays lost per exacerbation, reported in number of days per flare-up
Time Frame: During an URTI or flare-up during the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: days per flare-up
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
days per flare-up | 1.7 [0.9 to 2.5] | 1.0 [0.3 to 1.7]

15. Other Pre Specified Outcome: Percent of Participants With at Least 1 Exacerbation Requiring Rescue Oral Corticosteroids
Description: The percentage of participants with ≥1 reported asthma exacerbations requiring rescue oral corticosteroids
Time Frame: During the 7-month follow-up period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
percentage of participants | 42 | 61

16. Other Pre Specified Outcome: Duration of Asthma Symptoms During a Flare-up (Verbal Report)
Description: Group difference in the duration of asthma symptoms by verbal report.
Time Frame: During an URTI or flare-up during the 7-month follow-up period
Measure: Mean (95% Confidence Interval); unit: days/exacerbation
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 24 | 23
days/exacerbation | 7.4 [5.8 to 9.0] | 7.6 [5.1 to 10.0]

ADVERSE EVENTS:
Arm/Group | Placebo | Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/23
Other Adverse Events (participants affected / at risk) | 17/24 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Vitamin D (N=23)
peribronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — requin hospitalisation
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Vitamin D (N=23)
General (SOC) (General disorders) | 17 (29) | 13 (18) — Includes: FEVER, FATIGUE, PAIN IN BOTH LEGS, PAIN LEFT HAND, TOOTHACHE, SLEEP DISORDER
infections and infestations (SOC) (Infections and infestations) | 17 (49) | 19 (39) — Includes: OTITIS, PNEUMONIA, PHARYNGITIS, GASTROENTERITIS, STREPTOCOCCUS PHARYNGITIS, SINUSITIS, CONJONCTIVITIS etc.
Respiratory (SOC) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) — Includes: BRONCHITIS/BRONCHIOLITIS, COUGH, ADENOID HYPERTROPHY, CHRONIC RHINITIS, SNEEZING
Blood and lymphatic system disorders (SOC) (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — Includes: HETEROZYGOTIE AC, ANEMIA, EPISTAXIS, SPLENOMEGALY
Ear and labyrinth disorders (SOC) (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Includes: Otalgia , Ruptured tympanic membrane
Eye disorders (SOC) (Eye disorders) | 1 (1) | 0 (0) — Strabism
Gastrointestinal disorders (SOC) (Gastrointestinal disorders) | 8 (11) | 3 (4) — Includes: VOMITING, CONSTIPATION, DIARRHEA, RECTAL PROLAPSUS
Immune system disorders (SOC) (Immune system disorders) | 5 (6) | 2 (3) — Allergy
Investigations (SOC) (Investigations) | 9 (16) | 7 (12) — Includes: ELEVATED CA:CR RATIO, INCREASE BLOOD PHOSPHORUS, LOW ALP, INCREASE IN BLOOD CALCIUM
Musculoskeletal disorders (SOC) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — PULLED ELBOW
Nervous system disorder (SOC) (Nervous system disorders) | 1 (1) | 1 (1) — Includes: SEIZURE, PERVASIVE DEVELOPMENT DISORDERS
Reproductive system (SOC) (Reproductive system and breast disorders) | 0 (0) | 1 (1) — PHIMOSIS
Skin and subcutaneous tissue disorders (SOC) (Skin and subcutaneous tissue disorders) | 4 (5) | 7 (10) — Includes: RASH/ERYTHEMA, ECZEMA, GIANOTTI CROSTI SYNDROME, LÉSIONS
Surgical and medical procedures (SOC) (Surgical and medical procedures) | 1 (1) | 1 (1) — Includes: FACE TRAUMA TEETH EXTRACTION, MYRINGOTOMY AND TUBE PLACEMENT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No